CLINICAL TRIAL: NCT07157085
Title: AI-Driven Multitask Model for Guiding Treatment Decision-Making in Hepatocellular Carcinoma
Brief Title: AI Multitask Model for HCC Treatment
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Wei Peng, Professor, Sun Yat-sen University
Other Study IDs: [2024]593
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC; artificial intelligence; multitask deep learning; clinical decision support
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Diagnostic liver biopsy specimens and postoperative surgical specimens obtained from the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comprehensive treatment — Comprehensive HCC therapies include liver resection, TACE, HAIC, targeted therapy, immunotherapy and radiotherapy

SUMMARY:
We will integrate multi-modal cardiac data via an AI multitask framework to develop and validate concurrent models for liver function, treatment prognosis, and microvascular invasion (MVI) prediction in hepatocellular carcinoma. The resulting tool will be prospectively deployed to guide personalized surgical, TACE, and systemic therapy decisions.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years;
2. HCC diagnosed according to the European Association for the Study of the Liver/American Association for the Study of Liver Diseases criteria)
3. Eastern Cooperative Oncology Group performance status < 2;
4. Child-Pugh class A or B liver function;

Exclusion Criteria:

1. HCC combined with other malignancies;
2. missing image data during perioperative period;
3. lost to follow-up > 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC received comprehensive therapies such as liver resection, ablation, TACE, HAIC, targeted therapy, immunotherapy and radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 60 months
  from diagnosis of HCC to death or last follow-up

SECONDARY OUTCOMES:
Progression-free survival | 60 months
  from diagnosis of HCC to disease progression or last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No